CLINICAL TRIAL: NCT05411627
Title: A Pilot Study of Shockwave Therapy for Lower Extremity Spasticity in Persons With Genetically-Confirmed HSP
Brief Title: A Pilot Study of Shockwave Therapy in HSP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding issues
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Adam Tenforde, Physician, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000682
Record Dates: First submitted 2022-05-27; First posted 2022-06-09 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Pilot group of all 8 anticipated participants
  Interventions: Device: Shockwave Therapy

INTERVENTIONS:
Device: Shockwave Therapy — Participants will receive shockwave therapy once per week for three weeks.

SUMMARY:
This is a pilot study of the efficacy, safety, and tolerability of shockwave therapy for the treatment of spasticity in Hereditary Spastic Paraplegia.

DETAILED DESCRIPTION:
This is a pilot study investigating the efficacy, safety, and tolerability of Extracorporeal Shockwave Therapy (ESWT) for the treatment of lower-extremity spasticity in the setting of Hereditary Spastic Paraplegia (HSP). 8 participants will be treated with shockwave therapy targeting sites of maximal spasticity in the lower extremities for 3 sessions at a rate of once per week. Participants will fill out baseline questionnaires assessing their overall wellbeing and function prior to treatment session 1, and will complete follow-up questionnaires at visit 2, visit 3, a phone call within 7 days of visit 3, and 8 weeks after initial visit. Total time enrolled in the study will be 8 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18
2. Diagnosis of genetically-confirmed HSP
3. Score of 2, 3 or 4 on the PLSFRS walking question
4. 30 days stable dosages of oral spasticity medications prior to screening and throughout study participation
5. Able to come to site for treatment sessions
6. Able to understand all study procedures

Exclusion Criteria:

1. Diagnosis of any other neurological disorder that may impact gait
2. Lower motor neuron (LMN) disease or combined UMN and LMN
3. Non-ambulatory or requiring two-person assistance for any functional ambulation on most days
4. Less than 3 months of symptoms
5. Have received SWT within the past 3 months
6. Prior botulinum toxin injection within 3 months or planning to receive botulinum toxin injections during the study participation for spasticity management
7. Presence of an intra-thecal baclofen pump
8. Women who are pregnant. This is due to the fact that pregnancy will reduce participants activity after the treatment and the safety concerns related to shockwave treatment.
9. Patients with neuropathy affecting sensation to pain
10. Patients with a known underlying cardiac disease that could be affected by shockwave therapy
11. Concomitant intake of another clinical trial or other off-label experimental treatments that might influence study outcomes
12. Presence of unstable psychiatric disease, cognitive impairments, or dementia impairing study participation
13. Presence of other chronic neurological diseases such as Alzheimer's Parkinson's, stroke, or multiple sclerosis
14. Personal history of narcotic overuse for chronic pain or substance abuse or dependence
15. Contraindications for ESWT, including local skin breakdown, infection, malignancy or other soft tissue pathology at sites of planned treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale for Pain | 0-8 weeks; assessed at baseline visit, 1, 2, 3, and 8 weeks
  A rating of pain from 0 (none) to 10 (worst)
Primary Lateral Sclerosis Functional Rating Scale (PLSFRS) | 0-8 weeks; assessed at baseline visit, 1, 3, and 8 weeks
  The score of the rating scale ranges from 0-68, where 68 is a person who is completely asymptomatic.
Neurological Quality of Life (Neuro-QoL) Questionnaire: Fatigue Short Form | 0-8 weeks; assessed at baseline visit, 1, 3, and 8 weeks
  The score of this questionnaire ranges from 8 (least fatigue) to 40 (most fatigue)
Foot and Ankle Ability Measure (FAAM) Questionnaire: Activities of Daily Living Subscale | 0-8 weeks; assessed at baseline visit, 1, 3, and 8 weeks
  The score of this questionnaire ranges from 0 (maximally symptomatic in activities of daily living) to 84 (asymptomatic in activities of daily living).
Global Rate of Change (GROC) Questionnaire | 0-8 weeks; assessed at baseline visit, 1, 3, and 8 weeks
  The score ranges from -7 (maximally negative change) to +7 (maximally positive change)
Neurological Quality of Life (Neuro-QoL) Questionnaire: Lower Extremity Function - Mobility Short Form | 0-8 weeks; assessed at baseline visit, 1, 3, and 8 weeks
  The score of this questionnaire ranges from 8 (minimal lower extremity function) to 40 (maximal lower extremity function)
Neurological Quality of Life (Neuro-QoL) Questionnaire: Positive Affect and Wellbeing Short Form | 0-8 weeks; assessed at baseline visit, 1, 3, and 8 weeks
  The score of this questionnaire ranges from 9 (minimal wellbeing) to 45 (maximal wellbeing)
Neurological Quality of Life (Neuro-QoL) Questionnaire: Satisfaction with Social Roles and Activities Short Form | 0-8 weeks; assessed at baseline visit, 1, 3, and 8 weeks
  The score of this questionnaire ranges from 8 (minimal satisfaction) to 40 (maximal satisfaction)
Foot and Ankle Ability Measure (FAAM) Questionnaire: Sports Subscale | 0-8 weeks; assessed at baseline visit, 1, 3, and 8 weeks
  The score of this questionnaire ranges from 0 (maximally symptomatic in sports activities) to 32 (asymptomatic in sports activities)
Ten-Meter Walk Test | 0-3 weeks; assessed at baseline visit, 1, 2, and 3 weeks
  Participants will be asked to walk ten meters 2x at their self-selected walking speed and 2x at their fast walking speed. Time taken to complete walks will be measured.

IPD SHARING:
Plan to Share IPD: No